CLINICAL TRIAL: NCT00147914
Title: A Comparison Study Between Cefdinir and Amoxicilline/Clavulanate in Patients With Acute Sinusitis and Assessment of Quality of Life (QOL)
Brief Title: Comparison Study Between Cefdinir & Amoxicilline/Clavulanate in Acute Sinusitis and Assessment of Quality of Life
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 11791A
Record Dates: First submitted 2005-09-02; First posted 2005-09-07 (Estimated); Last update posted 2017-05-02 (Actual); Status verified 2017-05

CONDITIONS: Acute Bacterial Sinusitis
Keywords: Acute bacterial sinusitis
MeSH Terms: interventions — Cefdinir; Pharmaceutical Preparations; Amoxicillin-Potassium Clavulanate Combination

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): cefdinir
  Interventions: Drug: Cefdinir (drug)
- 2 (Active Comparator): amoxicillin/clavulanate
  Interventions: Drug: amoxicillin/clavulanate

INTERVENTIONS:
Drug: Cefdinir (drug) — cefdinir 300mg per orally twice daily for 10 days
  Arms: 1
Drug: amoxicillin/clavulanate — 1000mg /62.5mg extended release per orally twice daily for 10 days
  Arms: 2

SUMMARY:
This study is a comparison between two commonly used antibiotics (Cefdinir vs. Amoxicillin/Clavulanate) in patients with acute sinus infection, surveying quality of life. The hypothesis is that the two treatments would be at the least equivalent based on clinical outcome measures of improvement in quality of life.

DETAILED DESCRIPTION:
The purpose if this investigation is to evaluate the rate of improvement ub Quality of LIfe (QOL) in two different medications, a 10-day course of Cefdinir 300 mg PO BID versus a 10-day course of Amoxicillin/Clavulanate 1000 mg/62.5 mg XR BID, in the treatment of acute bacterial sinusitis.

ELIGIBILITY:
Inclusion Criteria:

* Male and female outpatient adults greater than 18 years old fulfilling the case definition for acute bacterial sinusitis
* Case definition includes clinical signs and symptoms, radiographic findings and collection of purulent material from the sinus

Exclusion Criteria:

* Symptoms less than 7 days and more than 3 weeks
* History of sinus surgery within 3 months
* History of frequent sinus infections (more than 2 episodes within the last 6 months)
* History of kidney and liver disease
* Pregnant and nursing women
* Pre-existing disease that could predispose to sinus infections (cystic fibrosis or nasal polyps
* Immunosuppressed patients
* History of allergy to either drug. Patients with a documented history of allergies to either penicillin or cephalosporins will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2005-02; Primary Completion 2007-02 (Actual); Study Completion 2017-02-18 (Actual)

PRIMARY OUTCOMES:
Improvement in quality of life | At baseline and within 1 week of completing treatment
SNOT 20 questionnaire | At baseline and within 1 week of completing treatment

SECONDARY OUTCOMES:
Clinical signs and symptoms alleviated | At baseline and within 1 week of completing treatment

CONTACTS AND LOCATIONS:
Overall Officials: Jacquelynne Corey, M.D., Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States

REFERENCES:
- [Background] Tantilipikorn P, Fritz M, Tanabodee J, Lanza DC, Kennedy DW. A comparison of endoscopic culture techniques for chronic rhinosinusitis. Am J Rhinol. 2002 Sep-Oct;16(5):255-60. PMID 12422969
- [Background] Vaidya AM, Chow JM, Stankiewicz JA, Young MR, Mathews HL. Correlation of middle meatal and maxillary sinus cultures in acute maxillary sinusitis. Am J Rhinol. 1997 Mar-Apr;11(2):139-43. doi: 10.2500/105065897782537133. PMID 9129756